CLINICAL TRIAL: NCT04885738
Title: The Value of Exhaled Nitric Oxide in Predicting Airway Eosinophilic Inflammation in Chronic Airway Inflammatory Disease
Brief Title: The Value of FeNO in Predicting Airway Eosinophilic Inflammation
Acronym: FeNO-Eos
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Huizhou Third People's Hospital (Unknown); Tongji Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Ruijin Hospital (Other); First Hospital of China Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Henan Provincial People's Hospital (Other); The Second Hospital of Hebei Medical University (Other); West China Hospital (Other); The First People's Hospital of Yunnan (Other); Inner Mongolia People's Hospital (Other); Second Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Kefang Lai, Professor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: FeNO-Eos
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Biomarkers; Airway Inflammation
MeSH Terms: interventions — Guidelines as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Cough: cough as a sole presenting lasted more than 8 weeks; with an age of 18-70years; with a normal chest X-ray; without steroids treatment in the last 4 weeks.
  Interventions: Other: no intervention
- Asthma: classic asthma
  Interventions: Other: no intervention
- COPD: patients with COPD in stable stage or acute exacerbation
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — For Chronic Cough，follow《Guidelines for the diagnosis and treatment of cough》(2015).
  For Asthma, follow GINA For COPD, follow GOLD.
  Other Names: guideline

SUMMARY:
To investigate and compare the value of FeNO, blood Eos, serum TIgE in predicting the airway eosinophilic inflammationin chronic cough, asthma and COPD.

DETAILED DESCRIPTION:
Cough is the most common complaint in the respiratory department, while asthma and chronic obstructive pulmonary disease(COPD) are two major respiratory disease that seriously endanger human health. The common test to identify the cause and evaluate the therapeutic effect such as induced sputum, pulmonary ventilation function test, bronchial provocation test, etc. are time-consuming and laborious. There is an urgent need for an easily detectable index in the clinic to quickly identify airway eosinophilic inflammation in chronic cough, asthma and COPD, which will provide important guidance for clinical treatment.

As a new marker of airway inflammation, exhaled nitric oxide(FeNO) can reflect eosinophilic airway inflammation. Mean while, FeNO has the advantages of non-invasive, simple operation, time-saving, labor-saving, and good reproducibility, which is suitable for clinical application.

This prospective, multi-center study aims to explore the value of FeNO in predicting airway eosinophilic inflammation and compare it with blood Eos and TLgE in patients with chronic cough, asthma and COPD.

ELIGIBILITY:
Inclusion Criteria:

* Candidates voluntarily participate in and abide by the relevant regulations of the study, can cooperate with corresponding inspections, follow the follow-up plan, and voluntarily sign written informed consent.
* Patients with chronic cough

  1. Coughing lasting ≥ 8 weeks,
  2. There is no obvious abnormality in the chest X-ray
  3. No clear history of upper respiratory tract infection in the past 4 weeks,
  4. Newly diagnosed or untreated in the last 4 weeks
  5. Non-smokers.
* Patients with Asthma

  1. For newly diagnosed and previously diagnosed asthma patients, the diagnosis criteria for asthma:
  2. Including various disease severity (mild, moderate, severe), various disease states (chronic duration, acute exacerbation period).
  3. Non-smokers.
* Patients with COPD 1) Including patients in stable phase and acute exacerbation phase.

Exclusion Criteria:

* Diagnose patients with ACO;
* Those who cannot cooperate with the completion of research-related test, follow-ups and other reasons cannot cooperate with the progress of the research;
* Combined with serious diseases of other systems (such as cardiovascular, metabolic, immune, neurological, etc.). With other diseases of the lung, including bronchiectasis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic cough, asthma, and COPD patients
Sampling Method: Probability Sample
Enrollment: 2052 (Estimated)
Dates: Start 2021-05-25 (Estimated); Primary Completion 2022-03-25 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
predictive value of FeNO in eosinophilic airway inflammation | 12 months
  predictive value of FeNO in eosinophilic airway inflammation in patients with chronic cough, classic asthma, COPD
predictive value of blood eosinophils in eosinophilic airway inflammation | 12 months
  predictive value of blood eosinophils in eosinophilic airway inflammation in patients with chronic cough, classic asthma, COPD
predictive value of TIgE in eosinophilic airway inflammation | 12 months
  predictive value of TIgE in eosinophilic airway inflammation in patients with chronic cough, classic asthma, COPD

SECONDARY OUTCOMES:
comparison of FeNO, blood eosinophils, TIgE in predicting eosinophilic airway inflammation | 12 months
  comparison the predictive value of FeNO, blood eosinophils, TIgE in eosinophilic airway inflammation in patients with chronic cough, classic asthma, COPD respectively
combination of biomarkers in predicting eosinophilic airway inflammation | 12 months
  combination of FeNO, blood eosinophils, TIgE in predicting eosinophilic airway inflammation in patients with chronic cough, classic asthma and COPD respectively

OTHER OUTCOMES:
correlation | 12 months
  correlation between FeNO and sputum eosinophils before and after the treatment in patients with chronic cough, asthma

CONTACTS AND LOCATIONS:
Overall Officials: Kefang Lai, phD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou Institute of Respiratory health, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Yi F, Chen R, Luo W, Xu D, Han L, Liu B, Jiang S, Chen Q, Lai K. Validity of Fractional Exhaled Nitric Oxide in Diagnosis of Corticosteroid-Responsive Cough. Chest. 2016 Apr;149(4):1042-51. doi: 10.1016/j.chest.2016.01.006. Epub 2016 Jan 22. PMID 26836931
- [Background] Lai K, Chen R, Lin J, Huang K, Shen H, Kong L, Zhou X, Luo Z, Yang L, Wen F, Zhong N. A prospective, multicenter survey on causes of chronic cough in China. Chest. 2013 Mar;143(3):613-620. doi: 10.1378/chest.12-0441. PMID 23238526
- [Background] Lane C, Knight D, Burgess S, Franklin P, Horak F, Legg J, Moeller A, Stick S. Epithelial inducible nitric oxide synthase activity is the major determinant of nitric oxide concentration in exhaled breath. Thorax. 2004 Sep;59(9):757-60. doi: 10.1136/thx.2003.014894. PMID 15333851
- [Background] Alving K, Malinovschi A. Basic aspects of exhaled nitric oxide. European Respiratory Monograph. 2010;49:1-31.
- [Background] Oh MJ, Lee JY, Lee BJ, Choi DC. Exhaled nitric oxide measurement is useful for the exclusion of nonasthmatic eosinophilic bronchitis in patients with chronic cough. Chest. 2008 Nov;134(5):990-995. doi: 10.1378/chest.07-2541. Epub 2008 Jun 26. PMID 18583518
- [Background] Sato S, Saito J, Sato Y, Ishii T, Xintao W, Tanino Y, Ishida T, Munakata M. Clinical usefulness of fractional exhaled nitric oxide for diagnosing prolonged cough. Respir Med. 2008 Oct;102(10):1452-9. doi: 10.1016/j.rmed.2008.04.018. Epub 2008 Jul 9. PMID 18614345
- [Background] Prieto L, Ferrer A, Ponce S, Palop J, Marin J. Exhaled nitric oxide measurement is not useful for predicting the response to inhaled corticosteroids in subjects with chronic cough. Chest. 2009 Sep;136(3):816-822. doi: 10.1378/chest.08-2942. Epub 2009 May 1. PMID 19411296
- [Background] Smith AD, Cowan JO, Filsell S, McLachlan C, Monti-Sheehan G, Jackson P, Taylor DR. Diagnosing asthma: comparisons between exhaled nitric oxide measurements and conventional tests. Am J Respir Crit Care Med. 2004 Feb 15;169(4):473-8. doi: 10.1164/rccm.200310-1376OC. Epub 2003 Nov 25. PMID 14644933
- [Background] Berry MA, Shaw DE, Green RH, Brightling CE, Wardlaw AJ, Pavord ID. The use of exhaled nitric oxide concentration to identify eosinophilic airway inflammation: an observational study in adults with asthma. Clin Exp Allergy. 2005 Sep;35(9):1175-9. doi: 10.1111/j.1365-2222.2005.02314.x. PMID 16164444
- [Background] Silkoff PE, Lent AM, Busacker AA, Katial RK, Balzar S, Strand M, Wenzel SE. Exhaled nitric oxide identifies the persistent eosinophilic phenotype in severe refractory asthma. J Allergy Clin Immunol. 2005 Dec;116(6):1249-55. doi: 10.1016/j.jaci.2005.09.029. Epub 2005 Nov 8. PMID 16337453
- [Background] Fukuhara A, Saito J, Sato S, Sato Y, Nikaido T, Saito K, Fukuhara-Nakagawa N, Inokoshi Y, Ishii T, Tanino Y, Ishida T, Munakata M. Validation study of asthma screening criteria based on subjective symptoms and fractional exhaled nitric oxide. Ann Allergy Asthma Immunol. 2011 Dec;107(6):480-6. doi: 10.1016/j.anai.2011.09.002. Epub 2011 Oct 1. PMID 22123376
- [Background] Korevaar DA, Westerhof GA, Wang J, Cohen JF, Spijker R, Sterk PJ, Bel EH, Bossuyt PM. Diagnostic accuracy of minimally invasive markers for detection of airway eosinophilia in asthma: a systematic review and meta-analysis. Lancet Respir Med. 2015 Apr;3(4):290-300. doi: 10.1016/S2213-2600(15)00050-8. Epub 2015 Mar 20. PMID 25801413
- [Background] Donohue JF, Jain N. Exhaled nitric oxide to predict corticosteroid responsiveness and reduce asthma exacerbation rates. Respir Med. 2013 Jul;107(7):943-52. doi: 10.1016/j.rmed.2013.02.018. Epub 2013 Apr 17. PMID 23601567
- [Background] Schneider A, Schwarzbach J, Faderl B, Welker L, Karsch-Volk M, Jorres RA. FENO measurement and sputum analysis for diagnosing asthma in clinical practice. Respir Med. 2013 Feb;107(2):209-16. doi: 10.1016/j.rmed.2012.10.003. Epub 2012 Oct 27. PMID 23107283
- [Background] Jatakanon A, Lim S, Kharitonov SA, Chung KF, Barnes PJ. Correlation between exhaled nitric oxide, sputum eosinophils, and methacholine responsiveness in patients with mild asthma. Thorax. 1998 Feb;53(2):91-5. doi: 10.1136/thx.53.2.91. PMID 9624291
- [Background] Jones SL, Kittelson J, Cowan JO, Flannery EM, Hancox RJ, McLachlan CR, Taylor DR. The predictive value of exhaled nitric oxide measurements in assessing changes in asthma control. Am J Respir Crit Care Med. 2001 Sep 1;164(5):738-43. doi: 10.1164/ajrccm.164.5.2012125. PMID 11549525
- [Background] Schleich FN, Seidel L, Sele J, Manise M, Quaedvlieg V, Michils A, Louis R. Exhaled nitric oxide thresholds associated with a sputum eosinophil count >/=3% in a cohort of unselected patients with asthma. Thorax. 2010 Dec;65(12):1039-44. doi: 10.1136/thx.2009.124925. Epub 2010 Jul 29. PMID 20671307
- [Background] Zhang YM, Lin JT. [The values of fractional exhaled nitric oxide in the diagnosis and treatment of chronic cough]. Zhonghua Jie He He Hu Xi Za Zhi. 2011 Jul;34(7):504-8. Chinese. PMID 22041775
- [Background] Lemiere C, Ernst P, Olivenstein R, Yamauchi Y, Govindaraju K, Ludwig MS, Martin JG, Hamid Q. Airway inflammation assessed by invasive and noninvasive means in severe asthma: eosinophilic and noneosinophilic phenotypes. J Allergy Clin Immunol. 2006 Nov;118(5):1033-9. doi: 10.1016/j.jaci.2006.08.003. Epub 2006 Sep 25. PMID 17088126
- [Background] Dweik RA, Boggs PB, Erzurum SC, Irvin CG, Leigh MW, Lundberg JO, Olin AC, Plummer AL, Taylor DR; American Thoracic Society Committee on Interpretation of Exhaled Nitric Oxide Levels (FENO) for Clinical Applications. An official ATS clinical practice guideline: interpretation of exhaled nitric oxide levels (FENO) for clinical applications. Am J Respir Crit Care Med. 2011 Sep 1;184(5):602-15. doi: 10.1164/rccm.9120-11ST. PMID 21885636
- [Background] ten Brinke A, Zwinderman AH, Sterk PJ, Rabe KF, Bel EH. Factors associated with persistent airflow limitation in severe asthma. Am J Respir Crit Care Med. 2001 Sep 1;164(5):744-8. doi: 10.1164/ajrccm.164.5.2011026. PMID 11549526
- [Background] Meijer RJ, Postma DS, Kauffman HF, Arends LR, Koeter GH, Kerstjens HA. Accuracy of eosinophils and eosinophil cationic protein to predict steroid improvement in asthma. Clin Exp Allergy. 2002 Jul;32(7):1096-103. doi: 10.1046/j.1365-2222.2002.01412.x. PMID 12100060
- [Background] Hastie AT, Moore WC, Li H, Rector BM, Ortega VE, Pascual RM, Peters SP, Meyers DA, Bleecker ER; National Heart, Lung, and Blood Institute's Severe Asthma Research Program. Biomarker surrogates do not accurately predict sputum eosinophil and neutrophil percentages in asthmatic subjects. J Allergy Clin Immunol. 2013 Jul;132(1):72-80. doi: 10.1016/j.jaci.2013.03.044. Epub 2013 May 21. PMID 23706399
- [Background] Westerhof GA, Korevaar DA, Amelink M, de Nijs SB, de Groot JC, Wang J, Weersink EJ, ten Brinke A, Bossuyt PM, Bel EH. Biomarkers to identify sputum eosinophilia in different adult asthma phenotypes. Eur Respir J. 2015 Sep;46(3):688-96. doi: 10.1183/09031936.00012415. Epub 2015 Jun 25. PMID 26113672
- [Background] Pacheco A, Faro V, Cobeta I, Royuela A, Molyneux I, Morice AH. Gastro-oesophageal reflux, eosinophilic airway inflammation and chronic cough. Respirology. 2011 Aug;16(6):994-9. doi: 10.1111/j.1440-1843.2011.02010.x. PMID 21651646
- [Background] Saha S, Brightling CE. Eosinophilic airway inflammation in COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(1):39-47. doi: 10.2147/copd.2006.1.1.39. PMID 18046901
- [Background] Zietkowski Z, Kucharewicz I, Bodzenta-Lukaszyk A. The influence of inhaled corticosteroids on exhaled nitric oxide in stable chronic obstructive pulmonary disease. Respir Med. 2005 Jul;99(7):816-24. doi: 10.1016/j.rmed.2004.12.008. PMID 15939243
- [Background] Antus B, Barta I, Horvath I, Csiszer E. Relationship between exhaled nitric oxide and treatment response in COPD patients with exacerbations. Respirology. 2010 Apr;15(3):472-7. doi: 10.1111/j.1440-1843.2010.01711.x. Epub 2010 Feb 24. PMID 20210889
- [Background] Franklin PJ, Stick SM, Le Souef PN, Ayres JG, Turner SW. Measuring exhaled nitric oxide levels in adults: the importance of atopy and airway responsiveness. Chest. 2004 Nov;126(5):1540-5. doi: 10.1378/chest.126.5.1540. PMID 15539724
- [Background] Olin AC, Rosengren A, Thelle DS, Lissner L, Bake B, Toren K. Height, age, and atopy are associated with fraction of exhaled nitric oxide in a large adult general population sample. Chest. 2006 Nov;130(5):1319-25. doi: 10.1378/chest.130.5.1319. PMID 17099006
- [Background] Gelb AF, George SC, Camacho F, Fraser C, Flynn Taylor C, Shakkottai S. Increased nitric oxide concentrations in the small airway of older normal subjects. Chest. 2011 Feb;139(2):368-375. doi: 10.1378/chest.10-1157. Epub 2010 Aug 12. PMID 20705799
- [Background] Zetterquist W, Pedroletti C, Lundberg JO, Alving K. Salivary contribution to exhaled nitric oxide. Eur Respir J. 1999 Feb;13(2):327-33. doi: 10.1034/j.1399-3003.1999.13b18.x. PMID 10065676
- [Background] Deykin A, Halpern O, Massaro AF, Drazen JM, Israel E. Expired nitric oxide after bronchoprovocation and repeated spirometry in patients with asthma. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):769-75. doi: 10.1164/ajrccm.157.3.9707114. PMID 9517589
- [Background] Sanders SP, Proud D, Permutt S, Siekierski ES, Yachechko R, Liu MC. Role of nasal nitric oxide in the resolution of experimental rhinovirus infection. J Allergy Clin Immunol. 2004 Apr;113(4):697-702. doi: 10.1016/j.jaci.2004.01.755. PMID 15100676
- [Background] Petsky HL, Kynaston JA, McElrea M, Turner C, Isles A, Chang AB. Cough and exhaled nitric oxide levels: what happens with exercise? Front Pediatr. 2013 Oct 24;1:30. doi: 10.3389/fped.2013.00030. eCollection 2013. PMID 24400276
- [Background] Silkoff PE, McClean PA, Slutsky AS, Caramori M, Chapman KR, Gutierrez C, Zamel N. Exhaled nitric oxide and bronchial reactivity during and after inhaled beclomethasone in mild asthma. J Asthma. 1998;35(6):473-9. doi: 10.3109/02770909809071000. PMID 9751064